CLINICAL TRIAL: NCT05970783
Title: A Multicenter, Randomized, Double-blind, Dose-parallel, Placebo-controlled Phase III Clinical Trial to Evaluate the Efficacy and Safety of Jincaopian Tablets in Subjects with Chronic Pelvic Pain After Pelvic Inflammatory Disease
Brief Title: A Study of Jincaopian Tablets on Chronic Pelvic Pain After Pelvic Inflammatory Disease
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Beijing Konruns Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Z-JCP-T-Ⅲ-2021-BJKC-01
Record Dates: First submitted 2023-07-13; First posted 2023-08-01 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2024-10

CONDITIONS: Chronic Pelvic Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Jincaopian Tablets group (Experimental): Patients receive Jincaopian Tablets 0.6g/day for 12 weeks.
  Interventions: Drug: Jincaopian Tablets
- Placebo group (Placebo Comparator): Patients receive a placebo 0.6g/day for 12 weeks.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Jincaopian Tablets — Jincaopian Tablets 0.2g tid p.o.
  Other Names: ZY5301
  Arms: Jincaopian Tablets group
Other: Placebo — Placebo 0.2g tid p.o.
  Arms: Placebo group

SUMMARY:
The objective of this phase III trial to evaluate the efficacy and safety of Jincaopian Tablets in the treatment of subjects with chronic pelvic pain after pelvic inflammatory disease

DETAILED DESCRIPTION:
Chronic pelvic pain is the major sequela of pelvic inflammatory disease and it's a common, burdensome, and costly condition that disproportionately affects women. This multicenter, randomized, double-blind, dose-parallel, placebo-controlled phase III clinical trial is designed to evaluate the efficacy and safety of Jincaopian Tablets in the treatment of subjects with chronic pelvic pain after pelvic inflammatory disease. In this trial, 414 subjects were enrolled and randomized to either "Jincaopian Tablets" group, or the "placebo" group in a 2:1 ratio. The treatment period is 12 weeks and the follow-up period is 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Meet the diagnostic criteria for chronic pelvic pain sequelae of pelvic inflammatory disease;
* The average VAS score of pain in the week before enrollment is ≥4;
* The McCormack scale of physical signs at the time of enrollment is 4 to 12 points (including 4 points and 12 points);
* Women aged 18 to 50 (including 18 and 50) with a history of sexual life;
* Voluntarily participate in this clinical trial, give informed consent and sign the informed consent form.

Exclusion Criteria:

* Pelvic inflammatory disease (acute attack);
* Pregnant or lactating women, women of childbearing age who are unwilling to take effective measures to prevent pregnancy during the trial and within 6 months after the trial;
* Previously diagnosed with cervical intraepithelial neoplasia, primary/secondary dysmenorrhea, pelvic stasis syndrome and chronic pelvic pain caused by other non-pelvic inflammatory diseases;
* Complicated with specific vaginitis such as vulvovaginal candidiasis, trichomonas vaginitis, bacterial vaginosis;
* Gynecological tumors (maximum diameter of uterine fibroids greater than 3cm and submucosal fibroids), endometriosis, adenomyosis, acute cervicitis, tuberculous pelvic inflammatory disease, interstitial cystitis and other diseases related symptoms;
* Placement of intrauterine device in the past 3 months; absence of uterus and bilateral appendages;
* Received related treatment or took drugs with similar functions and indications within 14 days before the introduction;
* Liver function: ALT or AST>1.5 times the upper limit of normal value；Renal function：Scr>1.0 times the upper limit of normal value;
* Serum CA125 and erythrocyte sedimentation > 1.1 times the upper limit of normal value.
* Combined with serious cardiovascular, cerebrovascular, hematopoietic system and other serious diseases;
* Have an allergic history to the experimental drug;
* Have a long history of alcoholism or drug abuse;
* Intellectual disabilities or mental disorders;
* Participated in other clinical trials within the past 3 months;
* The investigator believes that it is not suitable to participate in this clinical trial.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 414 (Estimated)
Dates: Start 2022-11-08 (Actual); Primary Completion 2024-03-11 (Actual); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Pain disappearance rate after 12 weeks of treatment | 12 Weeks
  The pain disappearance referred to the Visual Analogue Scale (VAS) score becoming 0-1 points, and was no longer greater than or equal to 2 points at any subsequent evaluation. The pain disappearance rate was defined as the proportion of patients who achieved a pain disappearance after treatment.

SECONDARY OUTCOMES:
Pain disappearance rate after 4 and 8 weeks of treatment | 8 Weeks
  The pain disappearance referred to the Visual Analogue Scale (VAS) score becoming 0-1 points, and was no longer greater than or equal to 2 points at any subsequent evaluation. The pain disappearance rate was defined as the proportion of patients who achieved a pain disappearance after treatment.
Change of weekly average Visual Analogue Scale (VAS) score from baseline after 12 weeks of treatment | 12 Weeks
  Visual Analogue Scale (VAS) was used to evaluate pelvic pain degree. The VAS score ranged from 0 to 10, and a higher score represented greater pain intensity. The average VAS value for a week was calculated by dividing the sum of the scores for each day of the week by the number of days the score was recorded.
The area under the VAS score-time curve | 12 Weeks
  AUC under the curve to evaluating pain levels
McCormick Scale | 12 Weeks
  The McCormack scale was used to score the patient's physical signs. The total score is 36 points, rated from twelve aspects including uterine tenderness (divided into four quadrants), abdominal tenderness or rebound pain (divided into four quadrants), left or right adnexal tenderness, uterine tenderness, and cervical lifting and swinging pain. The scoring criteria was as following: no pain is 0 points; Mild pain without facial expression changes and muscle tension is 1 point; Pain accompanied by facial expressions and muscle tension is 2 points; Pain drama is 3 points.
General quality of life (Short Form-12) scale | 12 Weeks
  The Short Form-12 is an abbreviated version of the original 36-item QOL questionnaire. It comprises 12 items with a mental component summary (MCS) and a physical component summary (PCS). Possible scores for mental and physical health-related QOL subscales range from 0 to 100 points, and a higher score is interpreted as better QOL.
Disease efficacy evaluation | 12 Weeks
  Disease efficacy was determined based on the change of the clinical signs and symptoms.
  Based on the evaluation criteria, the Disease efficacy was recorded as Clinical recovery, significant effect, effectiveness, and ineffectiveness.
  Clinical recovery: The symptoms and signs disappear, and the integral values of symptoms, signs, and auxiliary examinations decrease by ≥ 95%.
  Significant effect: The symptoms and signs are significantly reduced, with a reduction of ≥ 70% and<95% in the score of symptoms, signs, and auxiliary examinations.
  Effective: Symptoms and signs have been alleviated, with a reduction of ≥ 30% and<70% in symptom, sign, and auxiliary examination scores.
  Invalid: No reduction or aggravation of symptoms and signs, with a decrease of<30% in the score of symptoms, signs, and auxiliary examinations
Adverse events (AEs) | 12 Weeks
  Incidence of treatment-related AEs

CONTACTS AND LOCATIONS:
Overall Officials: Xiuxiang Teng, Principal Investigator — Beijing Hospital of Traditional Chinese Medicine
Locations (1):
- Beijing Hospital of Traditional Chinese Medicine affiliated to Capital Medical University, Beijing, Beijing Municipality, China